CLINICAL TRIAL: NCT07094074
Title: Exploratory Functional Assessment After Lower Limb Amputation: Locomotion, Balance, Energy Performance and Strategies for Adapting to Orthopaedic Devices
Acronym: AMILOCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ORNETTI 2025
Record Dates: First submitted 2025-05-20; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lower Limb Amputation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No change of equipment at the inclusion visit (Experimental)
  Interventions: Other: Walk tests; Other: Functional testing; Other: Balance analysis; Other: Quantified analysis of walking; Other: Questionnaires
- Change of equipment at the end of the inclusion visit (Experimental)
  Interventions: Other: Walk tests; Other: Functional testing; Other: Balance analysis; Other: Quantified analysis of walking; Other: Questionnaires

INTERVENTIONS:
Other: Walk tests — * 200 m walk test
  * 2-minute walk test
  * 6-minute walk test
Other: Functional testing — Timed Up and Go test (TUG), Berg Balance Test (BBT), Choice Stepping Reaction Time (CSRT), Functional Reach Test (FRT)
Other: Balance analysis — Balance analysis
Other: Quantified analysis of walking — On flat ground, even on slopes and stairs
Other: Questionnaires — Houghton, Prosthetic Profile of the Amputees-Locomotion Capabilities Index (PPA-LCI), Activities-specific Balance Confidence scale (ABC), quality of life assessed by the SF-12

SUMMARY:
The general aim of this exploratory study is therefore to investigate and quantify the functional capacities of patients with lower limb amputations (transtibial and transfemoral), with no change in their management, and to describe any changes in these capacities. The volunteers included in this study will be testing new equipment, all of which will be CE-marked, and will therefore meet all the safety and performance conditions required for use by these patients (equipment that is likely to be prescribed as standard). These devices could benefit from current technological advances that could improve these patients' functional abilities. They will be chosen and adapted according to the volunteer's activity and current equipment.

This is a local project of the CHU Dijon Bourgogne which will take place on the Technological Investigation Platform located at the Centre de Rééducation et de Réadaptation of the CHU Dijon Bourgogne.

A maximum of 100 patients will take part in the study, divided into two sub-groups of between 5 and 50 patients, depending on the type of brace worn and the level of amputation.

After the inclusion visit, each volunteer will undergo 2 assessment visits (the order of assessment of the devices will depend on randomisation) separated by 3 to 6 weeks. Follow-up is for a maximum of 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent
* Patient able to understand simple commands and packaging instructions
* Male or female patient over 18 years of age
* Patient with a lower limb amputation, at tibial or femoral level

Exclusion Criteria:

* Person not affiliated to or not benefiting from a social security scheme
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a judicial protection measure
* Pregnant women, women in labour or breastfeeding mothers
* Adults who are incapable or unable to give their consent
* Subjects with disarticulated hips
* Subjects with serious associated pathologies having an impact on walking (other than amputation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Spontaneous walking speed before and after changing or modifying the equipment | Up to 14 weeks